CLINICAL TRIAL: NCT00435331
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study to Evaluate the Safety and Efficacy of 6R-BH4 in Subjects With Pulmonary Arterial Hypertension
Brief Title: 6R-BH4 Pulmonary Arterial Hypertension Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Ivan Robbins, Ivan Robbins, MD Professor of Medicine, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WILK1
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PPH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Open Label
  Interventions: Drug: sapropterin dihydrochloride (6R-BH4)

INTERVENTIONS:
Drug: sapropterin dihydrochloride (6R-BH4) — 2.5 mg/kg/day for two weeks, 5 mg/kg/day for two weeks, 10 mg/kg/day for four weeks, then 20 mg/kg/day for two days

SUMMARY:
The purpose of this study is to determine whether the addition of sapropterin dihydrochloride (6R-BH4) to existing treatment has any effect in patients with pulmonary arterial hypertension (PAH). Patients with PAH have low levels of a substance called nitric oxide (NO). Tetrahydrobiopterin (BH4) is a substance produced by the body that is an essential requirement in the formation of NO. NO is thought to be helpful in keeping blood vessels in the lung healthy. 6R-BH4 is an experimental (unproven) medicine made in the lab that is very much like the BH4 that our own body makes. The researchers are investigating whether 6R-BH4 can be added safely to current treatment for PAH and whether there is any evidence of benefit from its use. The study will take approximately one year to complete from the time recruitment begins.

The primary objective of the study is to evaluate the safety of oral 6R-BH4, administered in escalating doses in addition to standard care, in subjects with pulmonary arterial hypertension (PAH).

The secondary objective of the study is to evaluate change in biochemical markers of endothelial dysfunction and nitric oxide synthetase activity (coupled and uncoupled) in subjects with PAH receiving escalating doses of oral 6R-BH4 in addition to standard care.

The third objective of the study is to evaluate change in biomarkers of disease progression, 6-minute walk (6MW) distance, Borg dyspnea scores, and quality of life (QOL) measures in subjects with PAH receiving escalating doses of oral 6R-BH4 in addition to standard care.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety of oral 6R-BH4, administered in escalating doses in addition to standard care, in subjects with pulmonary arterial hypertension (PAH).

The secondary objective of the study is to evaluate change in biochemical markers of endothelial dysfunction and nitric oxide synthetase activity (coupled and uncoupled) in subjects with PAH receiving escalating doses of oral 6R-BH4 in addition to standard care.

The third objective of the study is to evaluate change in biomarkers of disease progression, 6-minute walk (6MW) distance, Borg dyspnea scores, and quality of life (QOL) measures in subjects with PAH receiving escalating doses of oral 6R-BH4 in addition to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of PAH, defined as mean pulmonary arterial pressure > 25 mm Hg (measured by catheter).
* PAH is primary (idiopathic) or is secondary and caused by collagen vascular disease, congenital heart disease, or thromboembolic disease.
* Modified New York Heart Association (NYHA) classification I, II, or III that has been stable for at least 8 weeks prior to enrollment.
* 6MW distance, as performed at screening or within three months (12 weeks) prior to screening, of ≥ 200 and ≤ 500 meters.
* Receiving stable doses of one or more medications that are approved for treatment of PAH, except for any agents specifically prohibited by this protocol, for a minimum of 12 consecutive weeks before enrollment. Note: anticoagulant therapy can be adjusted according to target INR.
* Receiving stable doses of concomitant medication for other conditions, except agents specifically prohibited by the protocol.
* At least 18 years of age and willing and able to complete an informed consent form.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study.

Exclusion Criteria:

* Previous treatment with any formulation of BH4.
* Known allergy or hypersensitivity to any excipient of 6R BH4.
* History of systemic hypotension, defined as systolic BP < 100 mm Hg and/or diastolic BP < 60 mm Hg.
* Treatment at screening or perceived need for treatment during the course of the study with any of the following:

  * intravenous epoprostenol
  * inhaled iloprost
  * subcutaneous treprostinil
  * levodopa
  * any PDE 3 inhibitor, such as cilostazol or milrinone
  * any drug known to inhibit folate metabolism, such as methotrexate (eg, TrexallR), tomizine, trimethoprim, sulfanilamide, deoxycoformycin
  * nitrates
* Diet supplementation with L-arginine or L-citrulline within 30 days of enrollment.
* Diet supplementation with high doses (> 3 times the recommended daily allowance) of antioxidants, such as Vitamin C.
* Use of any investigational product or device within 30 days prior to screening, or known requirement for any investigational agent prior to completion of all scheduled study assessments.
* Known to be positive for human immunodeficiency virus (HIV).
* An additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities. Concurrent disease or condition that may interfere with study participation or safety include bleeding disorders, arrhythmia, organ transplant (other than lung), organ failure, current neoplasm, poorly controlled diabetes mellitus, and serious neurological disorders.
* Serum creatinine > 2.0 mg/dL (180 μM/L) or hepatic enzyme levels more than 2 times the upper limit of normal.
* Pregnant or lactating at screening, or planning to become pregnant (self or partner) at any time during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of oral 6R-BH4, administered in escalating doses in addition to standard care, in subjects with pulmonary arterial hypertension (PAH). | Up to 14 weeks

SECONDARY OUTCOMES:
Change in biochemical markers of endothelial dysfunction and nitric oxide synthetase activity (coupled and uncoupled). | Up to 14 weeks
Change in biomarkers of disease progression, 6-minute walk (6MW) distance, Borg dyspnea scores, and quality of life (QOL) measures. | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ivan M. Robbins, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States